CLINICAL TRIAL: NCT05232266
Title: The Effectiveness of a Caralluma Fimbriata Extract on Stress, Sleep and Neurotransmitters, a Randomised Placebo-controlled Double-blind Study
Brief Title: The Effectiveness of a Caralluma Fimbriata Extract on Stress, Sleep and Neurotransmitters
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARSTA-21
Record Dates: First submitted 2022-01-18; First posted 2022-02-09 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Stress; Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caralluma fimbriata (Experimental): Caralluma fimbriata in capsule form - taken as a 500mg dose (two 250mg capsules) twice daily, morning and evening with food.
  Interventions: Drug: Caralluma Fimbriata
- Placebo comparator capsule - Microcrystalline cellulose (Placebo Comparator): A comparator capsule taken as a 500mg dose (two 250mg capsules) twice daily, morning and evening with food.
  Interventions: Drug: Placebo comparator - Microcrystalline cellulose

INTERVENTIONS:
Drug: Caralluma Fimbriata — Caralluma fimbriata in capsule form - taken as a 500mg dose (two 250mg capsules) twice daily, morning and evening with food.
  Other Names: C.fimbriata
  Arms: Caralluma fimbriata
Drug: Placebo comparator - Microcrystalline cellulose — Placebo comparator in capsule form - taken as a 500mg dose (two 250mg capsules) twice daily, morning and evening with food.
  Arms: Placebo comparator capsule - Microcrystalline cellulose

SUMMARY:
This is a double blind, randomised, placebo-controlled clinical trial aiming to assess the effectiveness of Caralluma fimbriata on stress, sleep and neurotransmitters in a healthy adult population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Self-reporting Stress
* Able to provide informed consent
* Agree not to change current diet and exercise program while enrolled in this trial
* Agree not to undertake another clinical trial while enrolled in this trial

Exclusion Criteria:

* Unstable or serious illness (e.g. Serious mood disorders, neurological disorders such as MS, kidney disease, liver disease, heart conditions, diabetes, thyroid gland dysfunction)*
* Current malignancy (excluding BCC) or chemotherapy and radiotherapy treatment for malignancy within the previous 2 years
* Receiving/prescribed coumadin (Warfarin), heparin, dalteparin, enoxaparin or other anticoagulation therapy
* Receiving treatment for anxiety, or taking supplements# for anxiety or sleep conditions such as saffron, valerian, etc.
* Active smokers, nicotine use, alcohol or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in the active or placebo formula
* Known pregnant or lactating woman
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other related clinical study during the past 1 month
* History of infection in the month prior to the study

  * An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

    * Potential participants that are taking supplements that would result in their exclusion must wait a 4-week washout period prior to commencing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Change in stress as assessed by Perceived Stress Scale (PSS) | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in stress as assessed by Perceived Stress Scale (PSS) - Score range 0-40, Higher scores indicate higher perceived stress.
Change in stress as assessed by Salivary Cortisol levels | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in stress as assessed by Salivary Cortisol levels through assay

SECONDARY OUTCOMES:
Change in stress and mood as assessed by the Profile of Mood States (POMS) scale | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in stress as assessed by Profile of Mood States (POMS) scale - Six dimensions including Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment assessed ona five point scale ranging from "not at all" to "extremely".
Change in stress and mood as assessed by The Depression, Anxiety Stress Scale -21 (DASS-21) | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in stress as assessed by DASS-21 - A set of three self-reported scales to measure emotional states of depression, anxiety and stress. Each scale contains 7 items.
Change in sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) which covers 7 domains with higher scores indicating poorer sleep quality.
Change in sleep as measured by the Restorative Sleep Questionnaire (RSQ) | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in sleep as assessed by the Restorative Sleep Questionnaire (RSQ) which has 9 items scaled from 1-5. Higher total scores indicate a more restorative sleep.
Change in Neurotransmitters as assessed by pathology | Baseline prior to commencement of study product, Week 4 and Week 8
  Change in neurotransmitters Serotonin, Dopamine, oxytocin, nor-epinephrine, adrenalin, glutamate and GABA as assessed by pathology

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Newstead, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared